CLINICAL TRIAL: NCT05453344
Title: DEXCOM ONE: Continuous Glucose Monitoring in the Real World, Utility of Sustained High Alerts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH22145
Record Dates: First submitted 2022-06-30; First posted 2022-07-12 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus
Keywords: Insulin-dependent
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention - DexCom one (Other): Provision of DexCom one for glucose monitoring
  Interventions: Device: DexCom one

INTERVENTIONS:
Device: DexCom one — Provision of DexCom One for glucose monitoring

SUMMARY:
The purpose of this study is to gather feedback on a new continuous glucose monitor (CGM), called DEXCOM One. Unlike some other CGMs which allow a low (hypoglycaemic) and a high (hyperglycaemic) glucose alarm to be set, the DEXCOM One sensor has the unique feature of the 'Sustained Hyperglycaemic Alert', where the alarm is only activated if the glucose is above a certain threshold for a pre-specified amount of time.

International consensus guidance states that people with diabetes should aim for 70% time in the range 3.9-10 mmol/L. After meals there is usually a rise in blood glucose, so it is not unexpected for the glucose to go above 10 mmol/L for a short time even if the insulin dose already given before a meal is correct. Therefore, people with a high glucose alarm set at 10 mmol/L on their GCM may unnecessarily inject extra insulin and risk a low blood glucose. However, DEXCOM One's Sustained Hyperglycaemic Alert would only notify patients if their blood sugar was high for a prolonged period, and so may reflect a time when it would be genuinely advantageous to inject more insulin.

The aim of this single-centre, non-randomised, observational study is to gather experience from a range of users to assess the utility of this unique attribute, and the optimal settings. We aim to recruit 80-100 patients, and each participant's involvement is in 2 phases; for the first 3 months DEXCOM One sensors will be used, and for months 4-6 there will be the option of continuing to use the DEXCOM One sensors with the addition of a FitBit to track physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+ years
* A patient registered in the diabetes service at Sheffield Teaching Hospitals NHS Foundation Trust
* HbA1c within the last 3 months of >70 mmol/mol

Exclusion Criteria:

* Unable to provide informed consent
* Unable to communicate in written and verbal English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months
  Change in venous HbA1c at 3 and 6 months compared to baseline

SECONDARY OUTCOMES:
rtCGM measurements | Baseline, 3 and 6 months
  Time glucose measurements are in range 3.9-10mmol/l, time above range 10-13.9, time significantly above range >14, time below range 3.0-3.8, and time significantly below range <3.0 mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Elliott, PhD, MbChB, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Teaching Hospital NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No